CLINICAL TRIAL: NCT04483518
Title: Epidemiological Survey of Hepatitis D Virus Infection in Hepatitis B Population Among Multi-center Hepatitis B Population in China
Brief Title: Epidemiological Survey of Hepatitis D Virus Infection in China
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); Shandong Provincial Hospital (Other Government); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Junqi Niu, Director of the department of Hepatology, The First Hospital of Jilin University
Other Study IDs: 19K056-001
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Observe and Describe the Prevalence of Hepatitis D Infection Among HBsAg Positive People
Keywords: HBsAg positive; HBV DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples are used to detect HDV antibodies or HDV RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBV patients: HBV patients with HBsAg positive and/or HBV DNA positive

SUMMARY:
This cross-sectional study will screen out hepatitis D virus-infected patients in HBsAg-positive people. Observe and describe the prevalence of hepatitis D infection among HBsAg positive people. The provinces of China are divided into 5 geographical areas (North, South, East, West and Central) to recruit patients according to the population density of each area. After statistical calculation, the total number of population needed is 3808.

DETAILED DESCRIPTION:
Entry criteria：1. Age 18 years and above. 2. male or female. 3. Diagnosed as chronic HBV infection (HBsAg positive) 4.Ability to sign informed consent.

Exclusion criteria：Patients who disagree to participate in the trial.

After the informed consent was signed, the quantitative data of the previous surface antigen or HBV DNA titer was collected during the return visit. 4 ml of venous blood was collected on the same day or the remaining serum from the surface antigen or hepatitis B quantitative test was collected for the detection of hepatitis D antibody and/or the quantitative detection of hepatitis D RNA.

After statistical analysis, calculate the hepatitis D infection status in China.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis B surface antigen or HBV DNA positive

Exclusion Criteria:

* Can't sign informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hepatitis B surface antigen or HBV DNA positive
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
The prevalence of hepatitis D virus | 2019-2020
  Proportion of hepatitis D infection in people with hepatitis B infection

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Dr., Study Director — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Infection rate data